CLINICAL TRIAL: NCT07206706
Title: Efficacy and Tolerability of Tadalafil 5mg Once Daily Versus Darifenacin for Ureteric Stent Related Symptoms
Brief Title: Efficacy and Tolerability of Tadalafil Versus Darifenacin in Management of Ureteric Stent-Related LUTS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MS221/2022
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2022-03

CONDITIONS: Management of Ureteric Stent Related LUTS and Pain
MeSH Terms: conditions — Pain | interventions — Tadalafil; darifenacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): in the 1st phase Group 1 received Tadalafil 5 mg tab once daily orally and switched to Darifenacin 7.5 mg once daily orally in the 2nd phase
  Interventions: Drug: Tadalafil 5Mg Tab; Drug: Darifenacin 7.5 MG
- Group 2 (Experimental): in the 1st phase: group 2 received darifenacin 7.5 mg once daily orally and switched to tadalafil 5 mg once daily orally in the 2nd phase of the study
  Interventions: Drug: Tadalafil 5Mg Tab; Drug: Darifenacin 7.5 MG

INTERVENTIONS:
Drug: Tadalafil 5Mg Tab — PDE5 inhibitor
Drug: Darifenacin 7.5 MG — anti muscarinic

SUMMARY:
This randomized, crossover clinical trial evaluated the efficacy and safety of tadalafil compared with darifenacin in managing lower urinary tract symptoms (LUTS) and pain related to indwelling ureteric stents. A total of 150 patients who underwent ureteric stent insertion after endoscopic treatment of ureteric stones were enrolled. Patients were randomized into two groups: Group 1 received tadalafil 5 mg once daily for 3 weeks, followed by a 1-week washout, then darifenacin 7.5 mg once daily for 3 weeks. Group 2 received the reverse sequence.

The primary outcome was change in LUTS as measured by a shortened International Prostate Symptom Score (IPSS). The secondary outcome was stent-related pain measured by the Numeric Pain Rating Scale (NPRS). Drug safety and tolerability were also assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-40 years
2. Patient with ureteric stent size 6 Fr-26 cm post endoscopic procedure.

Exclusion Criteria:

1. Known prostatic patient with LUTS
2. Pregnant or lactating women
3. Recurrent urinary tract infection.
4. Neurological diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
change in stent related lower urinary tract symptoms (LUTS) | 3 weeks
  Change from baseline in stent-related symptoms, measured by a shortened International Prostate Symptom Score (IPSS), including incomplete emptying (Q1) and storage domain (Q2, Q4, Q7). The score was calculated (minimum 0 and maximum 20) according to patients' answers to the questions Higher scores indicate worse symptoms.
Change in numerical Pain rating score (NPRS) | 3 weeks
  Change from baseline in ureteric stent-related pain, measured by the Numeric Pain Rating Scale (0 = no pain, 10 = worst pain).

SECONDARY OUTCOMES:
Incidence of Adverse Events | Throughout the 7-week study period (3 weeks first drug, 1 week washout, 3 weeks second drug)
  Number and type of drug-related adverse events (e.g., dry mouth, constipation, headache, flushing, myalgia), recorded during each treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: hossam M elawady, MD, Principal Investigator — urology department, Ain shams university
Locations (1):
- Ain Shams University Hospita, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the current study will not be publicly available due to institutional restrictions, but are available from the corresponding author on reasonable request.